CLINICAL TRIAL: NCT05117112
Title: Nutritional Biomarkers of Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 262590
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Three groups of subjects will be studied: young/health, older/healthy, and older/sarcopenic.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10g of nutritional product (Experimental): All subjects will ingest 10g of a commercially available nutritional supplement one time during a study visit.
  Interventions: Dietary Supplement: XS Muscle Multiplier

INTERVENTIONS:
Dietary Supplement: XS Muscle Multiplier — Distributed by Amway; this product is a powder, sold in a 6.8 ounce (192g) container.

SUMMARY:
This study proposes to characterize skeletal muscle amino acid kinetics to an EAA challenge, i.e., an oral amino acid tolerance test (OATT), in order to determine the state of muscle health. Analogous to the oral glucose tolerance test (OGTT) used to characterize alterations in glucose metabolism, the proposed OATT represents a potential low-cost solution to classifying patients' skeletal muscle health. The extrapolation of this work is the development of a simple analytical tool that would provide clinicians the ability to discern alterations in muscle amino acid kinetics prior to a loss of function.

DETAILED DESCRIPTION:
Sarcopenia increases the risk of a number of deleterious health conditions and represents a major financial cost to our healthcare system. Among older adults who are hospitalized, those with sarcopenia on admission are 5-fold more likely to incur higher hospital costs than those without. The operational definition of sarcopenia is defined as meeting the criteria for all of the following: low muscle strength, low muscle quantity or quality, and low physical performance. The diagnosis of sarcopenia requires techniques that are both expensive and operator-dependent. Simple measurements, such as BMI, do not necessarily identify sarcopenia. Importantly, current techniques can only identify sarcopenia after a physical/functional impairment has occurred. Skeletal muscle amino acid kinetics predict muscle health and functionality. Altered amino acid kinetics lead to decrements in muscle mass, quality, and performance. Muscle response to circulating essential amino acids (EAA) determines muscle amino acid kinetics. Thus, this study proposes to characterize skeletal muscle amino acid kinetics to an EAA challenge, i.e., an oral amino acid tolerance test (OATT), in order to determine the state of muscle health. Analogous to the oral glucose tolerance test (OGTT) used to characterize alterations in glucose metabolism, the proposed OATT represents a potential low-cost solution to classifying patients' skeletal muscle health. The extrapolation of this work is the development of a simple analytical tool that would provide clinicians the ability to discern alterations in muscle amino acid kinetics prior to a loss of function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 30 and 70-89 yrs

Exclusion Criteria:

* History of diabetes that requires insulin for control of blood glucose
* History of malignancy or chemo/radiation therapy in the 6 months prior to enrollment
* History of gastrointestinal bypass/reduction surgery (Lapband, gastric sleeve, etc.)
* Pregnant females
* Unwilling to wear the breath-collection mask
* Subjects who cannot refrain from using protein or amino acid supplements for 7 days prior to Visit 2
* Concomitant use of oral or injectable corticosteroids
* Concomitant use of testosterone, IGF-1, or similar anabolic agent
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Church, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Young: 18 to 30 years old.
- Healthy Elderly: Greater than or equal to 70 years of age. Handgrip greater than 35.5 and 20 for men and women, respectively.
- Sarcopenic Elderly: Greater than or equal to 70 years of age. Handgrip less than 35.5 and 20 for men and women, respectively.
Period: Overall Study
Arm/Group | Healthy Young | Healthy Elderly | Sarcopenic Elderly
Started | 9 | 11 | 10
Completed | 9 | 10 | 10
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Young | Healthy Elderly | Sarcopenic Elderly | Total
Number analyzed (Participants) | 9 | 10 | 10 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 0 | 0 | 9
  >=65 years | 0 | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (3.2) | 75.5 (5.5) | 77.1 (3.9) | 60.4 (23.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 4 | 21
  Male | 1 | 1 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 10 | 10 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Resting and Maximum Plasma Leucine Concentration
Description: The amount of leucine in the plasma at rest, following an overnight fast. Then maximum concentration of plasma leucine was the higher concentration observed following ingestion of the drink. The maximum amount can be different for everyone but typically occurs 45 to 75 minutes after consumption of the amino acid drink
Time Frame: A 5-hour period.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Healthy Young | Healthy Elderly | Sarcopenic Elderly
Number analyzed (Participants) | 9 | 10 | 9
micromoles per liter
  Max Plasma Leucine Concentration | 659 (128) | 755 (67) | 721 (114)
  Resting Plasma Leucine Concentration | 95 (21) | 100 (22) | 100 (21)

ADVERSE EVENTS:
Time Frame: From enrollment to the completion of the study day. Approximately 2 weeks.
Arm/Group | Healthy Young | Healthy Elderly | Sarcopenic Elderly
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT05117112/Prot_SAP_000.pdf